CLINICAL TRIAL: NCT02652221
Title: Determination of Liver Stiffness in Chronic Liver Disease Patients by Acoustic Radiation Force Imaging (ARFI) Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Siemens Medical Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-0478
Record Dates: First submitted 2016-01-04; First posted 2016-01-11 (Estimated); Results first posted 2017-07-12 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-06

CONDITIONS: Chronic Liver Disease
MeSH Terms: interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study cohort (Experimental): Acoustic Radiation Force Imaging
  Interventions: Device: Acoustic Radiation Force Imaging

INTERVENTIONS:
Device: Acoustic Radiation Force Imaging — ARFI US is a novel technique, recently FDA approved for use in children and adults, which provides an alternative method for quantifying liver stiffness.
  Other Names: ARFI

SUMMARY:
A prospective, pilot study using acoustic radiation force imaging (ARFI) ultrasound (US) to quantify liver stiffness in children and young adults with chronic liver disease. ARFI results will be compared to the current clinical standard of Magnetic Resonance Elastography (MRE) and to liver biopsy when available.

DETAILED DESCRIPTION:
ARFI US is a novel technique, recently FDA approved for use in children and adults, which provides an alternative method for quantifying liver stiffness. ARFI US has been shown in a small pilot investigation in Europe in children to be reliable and rapid in estimating moderate to severe liver stiffness using histology as a reference gold standard. ARFI measures the speed of a shear wave in the examined tissue, expressed in m/s. This shear wave velocity can be mathematically converted into a liver stiffness value, which can then be used to estimate degree of liver fibrosis. The technique is non-invasive, uses no ionizing radiation, and is fast (several minutes to complete). It is possible that ARFI US will be more accurate than MRE in quantifying liver stiffness. In addition, ARFI US will ultimately be a less expensive clinical test, shorter in duration, and will not require sedation/anesthesia in younger children as MRE requires.

ELIGIBILITY:
Inclusion Criteria:

* Less than 25 years old with chronic liver disease

Exclusion Criteria:

* Subjects without clinically ordered MRE
* Subjects who cannot cooperate with performance of the short ARFI exam

Ages: 1 Day to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 55 (Actual)
Dates: Start 2014-06; Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Trout, M.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study Cohort
Started | 55
Completed | 55
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Presenting for MR elastography
Arm/Group | Study Cohort
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 14 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 55
BMI [Mean (Standard Deviation); unit: kg/m2] | 29.1 (8.7)

OUTCOME MEASURES:

1. Primary Outcome: Agreement in Measured Liver Stiffness Between ARFI and MRE
Description: The investigators are seeking to define agreement between ARFI and MRE liver stiffness measurements obtained in the same patients on the same day to determine if the modalities can be used interchangeably for measurement of liver stiffness and prediction of significant liver fibrosis
Time Frame: Within 24 hours
Measure: Number; unit: kPa
Groups:
- BMI <30 kg/m2: Subset of study cohort with BMI <30 kg/m2
- BMI >30kg/m2: Subset of study cohort with BMI 30 kg/m2 or more
Arm/Group | BMI <30 kg/m2 | BMI >30kg/m2
Number analyzed (Participants) | 27 | 28
kPa
  Mean Stiffness by MRE | 3.21 | 2.48
  Mean Stiffness by ARFI | 1.81 | 2.0

2. Primary Outcome: Agreement in Measured Liver Stiffness Between ARFI and MRE
Description: as for outcome 1
Time Frame: Within 24 hours
Measure: Number; unit: Correlation Coefficient (rho)
Arm/Group | BMI <30 kg/m2 | BMI >30kg/m2
Number analyzed (Participants) | 27 | 28
Correlation Coefficient (rho) | 0.61 | 0.07

ADVERSE EVENTS:
Time Frame: Study period
Arm/Group | Study Cohort
All-Cause Mortality (participants affected / at risk) | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55
Other Adverse Events (participants affected / at risk) | 0/55

LIMITATIONS AND CAVEATS:
1)Did not compare ARFI from multiple vendors to MR elastography, 2)No histologic reference standard

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No